CLINICAL TRIAL: NCT05316545
Title: Retrospective Analysis of Anesthesia Procedure in Orthognathic Surgery
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-E(I)-20210262
Record Dates: First submitted 2022-01-10; First posted 2022-04-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2021-12

CONDITIONS: Orthognathic Surgery
Keywords: orthognathic surgery; anesthesia; retrospective analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Using retrospective medical records to analyze the difference between the analysis of the correlation between operation time, blood loss, anesthesia methods, anesthesia medication, and postoperative recovery time

DETAILED DESCRIPTION:
In Orthognathic surgery, facial bones involved in the operation site are more likely to bleed. In order to reduce the amount of bleeding during the operation, intentional hypotensive anesthesia is executed during the operation.

Because the amount of bleeding is controlled within a reasonable range, the surgical field of vision is naturally clear, which can also make the operation go smoothly, shorten the operation time, and increase the postoperative comfort. Therefore, for orthognathic surgery, the maintenance of intraoperative blood pressure is very important. Using inhaled anesthetics can easily achieve deeper anesthesia, but may increase postoperative nausea and vomiting. Generally speaking, these patients will be fixed with steel wires between the upper and lower jaws after the operation. Postoperative nausea and vomiting will increase the risk of aspiration pneumonia, but intravenous anesthesia can reduce postoperative nausea and vomiting.

This research is a retrospective investigation of medical records. The purpose of this study is to understand the differences in the analysis of the correlation between the operation time, blood loss, anesthesia method, anesthesia medication, and postoperative recovery of patients undergoing surgery during orthognathic surgery. In the future, orthognathic surgery (Orthognathic surgery) anesthesia policy and anesthesia target process guidelines can be formulated, and it can help remind medical staff to make an early and appropriate treatment at any time.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing conventional anesthesia surgery and orthognathic surgery.

Exclusion Criteria:

* Exclude the operation time greater than 8 hours.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Review the operation time, blood loss, anesthesia method, anesthesia medication, and postoperative recovery evaluation of the operation record sheet and anesthesia-related record sheet (including the recovery room and postoperative visit record sheet) in the patient's medical record.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
medical treatment events performed | During procedure
  The purpose of the study is to analyze the cases of orthognathic surgery in our hospital from 2010 to 2021 and find out which medical treatment events must be performed while maintaining Intentional hypotension such as inhaled anesthetics, pain relievers, Nitroglycerine, target controlled infusion, Precedex, Opioid, antagonist also the timing when the medical treatment intervene.

SECONDARY OUTCOMES:
time of anesthesia,lose of blood and recovery after surgery | During procedure
  The secondary outcome will be analyzed for whether the medical treatment event would affect the time of anesthesia and loose of blood during the operative, and recovery after surgery,etc. We will collect the following data from electronic medical records: age, gender, weight, height, body mass index (BMI), preoperative American Society of Anesthesiologists (ASA) score, duration of anesthesia, type of anesthesia, anesthetic drugs, operation time, types of operation, estimated intraoperative blood loss (EBL), preoperative and postoperative Hemoglobin (HGB) and hematocrit (HCT), as well as postoperative recovery and statistically analyze the data by t-test and one-way ANOVA to get the mean and standard deviation of them.

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-I Cheng, Phd, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Sanmin Dist, Taiwan